CLINICAL TRIAL: NCT06224660
Title: A Phase 1b, Open-Label, Controlled Trial Evaluating the Safety and Efficacy of SRD-001 (AAV1/SERCA2a) in Subjects With Cardiomyopathy Secondary to Duchenne Muscular Dystrophy
Brief Title: Modulation of SERCA2a of Intra-Myocytic Calcium Trafficking in Cardiomyopathy Secondary to Duchenne Muscular Dystrophy
Acronym: MUSIC-DMD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sardocor Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SRD-001-1004
Record Dates: First submitted 2024-01-11; First posted 2024-01-25 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: DMD-Associated Dilated Cardiomyopathy
MeSH Terms: conditions — Dmd-Associated Dilated Cardiomyopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): SRD-001
  Interventions: Genetic: SRD-001
- High Dose (Experimental): SRD-001
  Interventions: Genetic: SRD-001
- Control (No Intervention): No-Intervention Control

INTERVENTIONS:
Genetic: SRD-001 — SRD-001 is an adeno-associated virus serotype 1 (AAV1) based gene therapy designed to deliver a copy of the gene encoding the human sarcoplasmic/endoplasmic reticulum Ca(2+) ATPase 2a (SERCA2a). It is administered as a one-time intracoronary infusion.
  Other Names: AAV1/SSERCA2a
  Arms: High Dose; Low Dose

SUMMARY:
This research study is testing whether an experimental drug, called SRD-001, is safe and helps the weakened heart of patients with Duchenne muscular dystrophy (DMD) regain its ability to effectively pump blood to the rest of the body. SRD-001 is a form of gene therapy. The goal of SRD-001 gene therapy is to provide the heart muscle cells with extra copies of the SERCA2a gene so that they can produce more SERCA2a protein to help the heart muscle cells squeeze/contract better. Researchers will compare SRD-001 treated participants with no-treatment participants; all participants will continue to take their current heart medications. All participants will be followed very closely for 2 years and undergo cardiac magnetic resonance imaging of their heart at baseline, year 1 and year 2 along with assessment of upper limb function and lung function. After the 2 years of close follow-up, all participants will roll over into long-term follow-up where they will be called biannually for information on their current medical status.

DETAILED DESCRIPTION:
This phase 1b, multi-center, non-randomized, open-label, ascending dose escalation, no-intervention-control trial will assess the safety and explore the efficacy of SRD-001 administered as a one-time antegrade epicardial coronary artery infusion for the treatment of participants with cardiomyopathy secondary to DMD. SRD-001 is an AAV1 vector expressing the transgene for SERCA2a. Twelve participants will be assigned to either active treatment with SRD-001 or no-intervention based upon their neutralizing antibody status. The objectives of the trial are (1) to evaluate the safety of a one-time intracoronary administration of SRD-001 in participants with cardiomyopathy due to DMD; and (2) to explore the impact of SRD-001 on heart and skeletal muscle function and quality of life. After screening to determine eligibility, participants will be sequentially assigned to low dose SRD-001, high dose SRD-001 or no-intervention. Participants assigned to active treatment with SRD-001 will under cardiac catheterization and angiography just prior to the intracoronary infusion of SRD-001 and spend overnight int he hospital for observation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DMD with confirmatory genetic testing
* Cardiomyopathy with left ventricular scar in at least 3 of 16 segments
* Left ventricular ejection fraction < 40%
* Individualized, optimized cardiac medical therapy and glucocorticoid treatment for at least 12 months prior to enrollment
* Willing and able to provide informed consent

Exclusion Criteria:

* Abnormal blood pressure
* Non-DMD-related liver function test elevations
* Cystatin C ≥ 1.2 mg/L
* Thrombocytopenia
* Anemia
* Inadequate pulmonary function

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Rate of all-cause mortality | From Day 1 to Week 52 and Week 104
  Death
Rate and severity of related treatment-emergent adverse events | From Day 1 to Week 52 and Week 104
  Adverse events related to the investigational product or the administration procedure
Rate and severity of all treatment-emergent adverse events | From Day 1 to Week 52 and Week 104
  Adverse events
Rate of cell-mediated immune reaction | From Day 1 to Week 52
  Cell-mediated immune reaction as assessed by enzyme-linked immunosorbent spot (ELISpot)

SECONDARY OUTCOMES:
Change, including normal/abnormal shifts, in 12-lead electrocardiogram (ECG) | From Day 1 to Week 52 and Week 104
  Change in the heart's electrical activity
Change, including normal/abnormal shifts, in laboratory evaluations | From Day 1 to Week 52 and Week 104
  Hematology, serum chemistries, urinalysis, cardiac enzymes and anti-AAV1 antibodies

OTHER OUTCOMES:
Change in myocardium and left ventricular structure and function | From baseline to Week 52 and Week 104
  Assessed by cardiac magnetic resonance imaging with late gadolinium enhancement
Change in skeletal muscle function | From baseline to Week 52 and Week 104
  Assessed by PUL 2.0, grip strength, key and tip-to-tip pinch strength and elbow flexion strength
Change in pulmonary function | From baseline to Week 52 and Week 104
  Assessed by slow vital capacity, forced expiratory volume in 1 second, forced vital capacity, peak expiratory flow, maximum inspiratory pressure, maximum expiratory pressure, peak cough flow and inspiratory flow reserve
Change in quality of life | From baseline to Week 52 and Week 104
  Assessed by the Duchenne muscular dystrophy quality of life questionnaire

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No